CLINICAL TRIAL: NCT06195436
Title: Efficacy of Acceptance and Commitment Therapy on Serum GDF-15 Levels in Older Adults With and Without Depression: a Non-randomized Intervention Study
Acronym: ACT GDF-15
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Colima (Other)
Responsible Party: Principal Investigator, Miguel Huerta, PhD Md, Universidad de Colima
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT_GDF15
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Conceptual definition: "It is framed in a functional philosophical position, it is based on a new Theory of Language and Cognition; offers an alternative to traditional psychopathology: the functional dimension of Experiential Avoidance; and promotes basic research and controlled trials".
  Operational definition: Participants with and without depression will be assigned to two study groups; both groups will undergo Acceptance and Commitment Therapy based on the required guidelines for twelve weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: For ethical reasons, it is methodologically inappropriate to randomize the study groups, so the protocol will adhere to the TREND guidelines (Transparent Reports of Non-randomized Evaluations [for its acronym in English: Transparent reporting of reviews with nonrandomized Designs ]), which share several criteria with CONSORTs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy for people with depression (Active Comparator): Acceptance and Commitment Therapy for people with depression
  Interventions: Behavioral: Acceptance and Commitment Therapy for people with and without depression
- Acceptance and Commitment Therapy for people without depression. (Active Comparator)
  Interventions: Behavioral: Acceptance and Commitment Therapy for people with and without depression

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy for people with and without depression — Participants with and without depression will be assigned to two study groups; both groups will undergo Acceptance and Commitment Therapy based on the required guidelines for twelve weeks.

SUMMARY:
In a world where the population is aging, strategies are required that promote physical, social and mental health in these age groups. Depression associated with biological aging is evidenced by clinical findings and biological markers in the course of the disease (such is the case of the GDF-15). The presence of mental health disorders, such as depression, favors the risk of premature mortality (even 25 years less than the general population, even controlling for the suicide variable.

In addition, older adult patients with depression have a higher risk of presenting chronic diseases, immunological alterations, and neurocognitive disorders , favoring accelerated aging that contributes to a reduction in their intrinsic and functional capacities. (51) .

GDF -15 has been proposed as a pro-aging protein , specifically promoted by mitochondrial dysfunction, which in turn leads to accelerated aging through oxidative stress.

In addition, considering that mental health requires care through therapies with the necessary scientific evidence to have an impact on the mental and physical health of older adults, therefore , Acceptance and Commitment Therapy is proposed as a way to lead to healthy aging that promotes less oxidative stress derived from the same depression. Therefore, the purpose of this study is focused on demonstrating the efficacy of acceptance and commitment therapy implemented for twelve weeks in a group of older adults with and without depression, and evaluating it considering the serum levels of GDF- 15 .

DETAILED DESCRIPTION:
Research question:

What is the efficacy of the implementation of Acceptance and Commitment Therapy in a group modality for twelve weeks on the serum levels of GDF-15 in older adults with and without depression?

General objective:

To determine the effectiveness of the implementation of Acceptance and Commitment Therapy in a group mode for twelve weeks on the serum levels of GDF-15 in older adults with and without depression .

Specific objectives:

* To determine the severity of depressive symptoms in the elderly participants.
* To assess the serum levels of GDF-15 in the elderly participants.
* To compare the serum levels of GDF-15 before and after the implementation of Acceptance and Commitment Therapy for twelve weeks in older adults with and without depression.
* To compare the depressive symptoms before and after the implementation of the Acceptance and Commitment Therapy and the control group for twelve weeks.
* Evaluate the adherence to the interventions carried out on the study participants.
* To establish the influence of age, sex, comorbidities and socioeconomic level on the efficacy of acceptance and commitment therapy and the control group in the participants.

Study hypothesis:

Older adults with depression show a greater decrease in serum GDF-15 levels after the implementation of Acceptance and Commitment Therapy in a group mode when compared to the group without depression for twelve weeks.

Type of research and variables:

Study Design: Non-randomized intervention study.

• For ethical reasons, it is methodologically inappropriate to randomize the study groups, so the protocol will adhere to the TREND guidelines (Transparent Reports of Non-randomized Evaluations [for its acronym in English: Transparent reporting of reviews with nonrandomized Designs ]), which share several criteria with CONSORTs.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 60 years of age of any gender with at least nine years of studies.
* People belonging to the group of Retirees and Pensioners of the University of Colima AC
* People who wish to voluntarily participate in the study.
* People with and without depression.

Exclusion Criteria:

* People who are undergoing psychological treatment or who in the last 12 months have undergone some psychological therapy.
* People under drug treatment for depression.
* People with a score of less than 23 points in the assessment of the cognitive state by the Minimental .
* People with medical diagnosis of neurocognitive diseases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
GDF-15 | 12 weeks
  the serum levels resulting from the measurement with the ELISA technique with a specific Kit for GDF-15. The values will be presented through the difference before and after both study interventions in each participant (value after the intervention - value before the intervention).

IPD SHARING:
Plan to Share IPD: Undecided